CLINICAL TRIAL: NCT00742742
Title: The Effects of Walnut Supplement on Cardio-Metabolic Risk Factors in Patients With Metabolic Syndrome
Brief Title: Walnut Intervention on Metabolic Syndrome (WIMS)
Acronym: WIMS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: California Walnut Commission (Other)
Responsible Party: Principal Investigator, Xu Lin, Principal Investigator, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CWC-2008; KSCX1-YW-02
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Metabolic Syndrome X
Keywords: Walnut; Lipids; Blood Glucose
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Nutrition advice (accroding to AHA recommendation) + 30 grams/day supplement of walnuts,walnuts were incorpatated into bread that provided to the participants
  Interventions: Behavioral: healthy life style education
- B (Sham Comparator): Registed dietians give the advice for health lyfestyle
  Interventions: Behavioral: healthy life style education

INTERVENTIONS:
Behavioral: healthy life style education — healthy life style education
  Other Names: Dietians provided healthy lifestyle education accroding to; AHA recommendation

SUMMARY:
The purpose of this study is to determine whether a daily supplement of 30 grams of walnut is effective in the treatment of metabolic syndrome (MetS).

DETAILED DESCRIPTION:
Metabolic syndrome (MetS), a constellation of metabolic abnormalities including central obesity, dyslipidemia, elevated blood pressure and hyperglycemia, is associated with the development of type 2 diabetes and CVD. It has become one of the major public health challenges in China due to rapidly nutrition transition and the nature of obesity epidemic. Treatment of MetS in China is very important for the prevention of the epidemic of its consequences (such as CVD and type 2 diabetes).

Compelling evidence from recent human studies has demonstrated that diet and lifestyle modifications are effective means in MetS management. Walnut is a complex food source containing high amounts of polyunsaturated fatty acids (PUFA), as well as plant protein, Vitamin E and other substances that may have an impact on health. Therefore, the aim of this study is to investigate the effect of walnut supplementation on the management of MetS in adult Chinese men and women in a randomized, controlled clinical trial. A total of 200 participants with MetS (defined by NCEP-ATPⅢ criteria) will be randomly assigned to a walnut-supplemented diet (30 grams/day) or an isocaloric control diet for 12 weeks. Effects of walnut supplementation will be evaluated by measuring metabolic profile (BMI, blood pressure, total cholesterol, triglyceride, LDL-C and HDL-C, fasting glucose and insulin, HbA1C), inflammatory markers (CRP and IL-6), markers of endothelial function (E-selectin, ICAM-1 and VCAM-1), and fatty acid profile.

ELIGIBILITY:
Inclusion Criteria:

* With metabolic syndrome. Metabolic syndrome was defined based upon the updated National Cholesterol Education Program Adult Treatment Panel III criteria for Asian-Americans as presenting at least 3 of the following components: 1) waist circumference ≥ 90 cm for men or ≥ 80 cm for women; 2) triglycerides ≥1.7mmol/l; 3) HDL cholesterol <1.03 for men or <1.30 for women; 4) blood pressure ≥130/85 mmHg, or current use of antihypertentive medications; 5) fasting glucose ≥5.6mmol/l or previously diagnosed type 2 diabetes or on oral antidiabetic agents or insulin.
* Being able to comply with the specified feeding conditions
* Being able to eat walnuts
* Being between the ages of 35 and 60 years

Exclusion Criteria:

* Pregnancy or lactation
* Use of insulin
* Severe kidney disease
* Cardiovascular diseases, stroke, cancer and psychological disorders
* Walnut allergies or frequently eating walnuts or other nuts (>90 grams/week)
* Drug or alcohol abuse.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome status | 12 weeks

SECONDARY OUTCOMES:
Total cholesterol, triglyceride, LDL_C HDL-C, fasting glucose and insulin, HbA1C, blood pressure, CRP, IL-6, adiponectin, RBP4, E-selectin, ICAM-1, VCAM-1, and fatty acid profiles of the red blood cells. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, MD, PhD, Principal Investigator — Institute for Nutritional Sciecnes, Chinese Acadamy of Sciences
Locations (1):
- Institute for Nutritional Sciecnes, Chinese Acadamy of Sciences, Shanghai, China

REFERENCES:
- [Derived] Wu H, Pan A, Yu Z, Qi Q, Lu L, Zhang G, Yu D, Zong G, Zhou Y, Chen X, Tang L, Feng Y, Zhou H, Chen X, Li H, Demark-Wahnefried W, Hu FB, Lin X. Lifestyle counseling and supplementation with flaxseed or walnuts influence the management of metabolic syndrome. J Nutr. 2010 Nov;140(11):1937-42. doi: 10.3945/jn.110.126300. Epub 2010 Sep 8. PMID 20826632